CLINICAL TRIAL: NCT01122927
Title: A Long-term, Multicenter, Open-Label Study to Evaluate the Safety and Tolerability of Flexible-Dose Oral Aripiprazole (OPC-14597) as Maintenance Treatment in Adolescent Patients With Schizophrenia or Child and Adolescent Patients With Bipolar I Disorder, Manic or Mixed Episode With or Without Psychotic Features
Brief Title: Safety and Tolerability of Aripiprazole in Adolescents With Schizophrenia or Children and Adolescents With Bipolar I Disorder, Manic or Mixed Episode With or Without Psychotic Features.
Acronym: ATTAIN 267
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was terminated early as the objective of the Aripiprazole Pediatric Investigational Plan was met and provided 2 years of safety data.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31-09-267
Record Dates: First submitted 2010-05-06; First posted 2010-05-13 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Adolescent Schizophrenia; Child or Adolescent Bipolar I Disorder, Manic or Mixed Episode With or Without Psychotic Features
Keywords: schizophrenia; adolescent; bipolar
MeSH Terms: conditions — Mania; Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase 1 and Phase 2 (Experimental): Aripiprazole (2-mg, 5-mg, 10-mg, 15-mg, 20-mg, 25-mg or 30-mg)
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole (2-mg, 5-mg, 10-mg, 15-mg, 20-mg, 25-mg or 30-mg) pill taken orally once per day

SUMMARY:
This is an open-label study consisting of a screening period, a conversion/titration phase (Phase 1), an open-label treatment phase (Phase 2), and a follow-up period.

The study will enroll new subjects (hereafter referred as "de novo" subjects) with schizophrenia, or bipolar I disorder, manic or mixed episode with or without psychotic features, and rollover subjects with schizophrenia from 31-09-266 (hereafter referred to as "Study 266"). All de novo subjects must enter the screening period of the study. Subjects who are screened and are not required to go through Phase 1 will complete a Phase 2 baseline visit prior to their participation in Phase 2.

Study Design: Treatment, Single Group Assignment, Open Label, Active Control, Safety/Efficacy Study

ELIGIBILITY:
Inclusion Criteria:

* Subjects 13-17 years old (Schizophrenia); Subjects 10-17 years old (Bipolar manic or mixed episode)* [*Bulgaria will enroll Schizophrenia subjects only.]
* Subjects with a current diagnosis of schizophrenia, and a history of the illness (diagnosis or symptoms) for at least 6 months prior to screening (as per subject, family, or healthcare provider, or by previous medical records).
* Subjects with a current diagnosis of bipolar I disorder, manic or mixed episode with or without psychotic features (diagnosis or symptoms) experiencing symptoms for at least 1 week prior to screening. * [*These subjects will not be eligible to enroll in Bulgaria]
* Subjects who have shown previous response to antipsychotic treatment (other than clozapine) and are not resistant to treatment with other antipsychotics.
* Subjects who are currently being treated with oral antipsychotics other than clozapine, and are not resistant to treatment with other antipsychotics.
* Inpatient or outpatient status, with the exception of acute hospitalization due to psychiatric reasons at the time of screening or before Phase 2.

Exclusion Criteria:

* All subjects: diagnosis of schizoaffective disorder, autism, pervasive developmental disorder (PDD), OCD, or PTSD.
* Subjects with schizophrenia: a current major depressive episode.
* Subjects with bipolar manic or mixed episode: presenting with a clinical picture and/or history that is consistent with a diagnosis of bipolar II disorder or bipolar disorder not otherwise specified.
* Subjects with delirium, dementia, amnesia or other cognitive disorders; subjects with psychotic symptoms that are better accounted for by another general medical condition(s) or direct effect of a substance (i.e., medication, illicit drug use, etc.).
* Subjects with any neurological disorder, with the exception of Tourette's syndrome.
* Subjects experiencing major depressive episode at the time of screening other than subjects diagnosed with bipolar I disorder mixed episode.
* Subjects who are currently receiving clozapine or have received clozapine at any time in the past are ineligible for entry into the study.
* Subjects who meet the DSM-IV-TR criteria for substance dependence (including alcohol and benzodiazepines, but excluding caffeine and nicotine) within the past 180 days prior to screening.
* Subjects who have epilepsy, a history of seizures (except for a single childhood febrile seizure or post-traumatic seizure), or a history of severe head trauma or stroke, or have a history or current evidence of other unstable medical conditions.
* Subjects with a history of subclinical hypothyroidism (TSH ≥ 4.0 mIU/L), known hypothyroidism, or hyperthyroidism (unless the condition has been stabilized with medications for at least 90 days prior to entry into Phase 1 or Phase 2).
* Subjects who have a medical history of uncontrolled diabetes, labile or unstable diabetes (brittle diabetes), newly diagnosed diabetes, or clinically significant abnormal blood glucose levels (defined as fasting blood glucose ≥ 125 mg/dL).

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 524 (Actual)
Dates: Start 2010-07; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kohegyi, MD, Study Director — Otsuka Pharmaceutical Development and Commercialization, Inc.
Locations (95):
- United States (22):
  - Study Site, Dothan, Alabama
  - Study Site, Downey, California
  - Study Site, Miami, Florida
  - Study Site, Atlanta, Georgia
  - Study Site, Smyrna, Georgia
  - Study Site, Oak Brook, Illinois
  - Study Site, Wichita, Kansas
  - Study Site, Minneapolis, Minnesota
  - Study Site, Buffalo, New York
  - Study Site, Stony Brook, New York
  - Study Site, Chapel Hill, North Carolina
  - Study Site, Cincinnati, Ohio
  - Study Site, Cleveland, Ohio
  - Study Site, Oklahoma City, Oklahoma
  - Study Site, Philadelphia, Pennsylvania
  - Study Site, Houston, Texas
  - Study Site, San Antonio, Texas
  - Study Site, The Woodlands, Texas
  - Study Site, Richmond, Virginia
  - Study Site, Bellevue, Washington
  - Study Site, Bothell, Washington
  - Study Site, Milwaukee, Wisconsin
- Bulgaria (8):
  - Study Site, Burgas
  - Study Site, Pazardzhik
  - Study Site, Plovdiv
  - Study Site, Rousse
  - Study Site 2, Sofia
  - Study Site, Targovishte
  - Study Site 1, Varna
  - Study Site 2, Varna
- Croatia (3):
  - Study Site, Rijeka
  - Study Site 1, Zagreb
  - Study Site 2, Zagreb
- Hungary (3):
  - Study Site, Budapest
  - Study Site, Gyula
  - Study Site, Szeged
- India (17):
  - Study Site, Vijayawada, Andhra Pradesh
  - Study Site, Visakhapatnam, Andhra Pradesh
  - Study Site 1, Ahmedabad, Gujarat
  - Study Site 2, Ahmedabad, Gujarat
  - Study Site, Ahmedabad, Gujarat
  - Study Site, Maninagar, Ahmedabad, Gujarat
  - Study Site, Mangalore, Karnataka
  - Study Site, Calicut, Kerala
  - Study Site, Nashik, Maharashtra
  - Study Site, Ludhiana, Punjab
  - Study Site, Jaipur, Rajasthan
  - Study Site, Chennai, Tamil Nadu
  - Study Site, Maduri, Tamil Nadu
  - Study Site, Kanpur, Uttar Pradesh
  - Study Site, Lucknow, Uttar Pradesh
  - Study Site, Varanasi, Uttar Pradesh
  - Study Site, Guntur
- Study Site, Kuala Lumpur, Kuala Lumpur, Malaysia
- Philippines (4):
  - Study Site, Dasmariñas, Cavite
  - Study Site, Manila, National Capital Region
  - Study Site, Iloilo City
  - Study Site, Mandaluyong
- Poland (4):
  - Study Site, Bialystok
  - Study Site, Gdansk Wrzeszcz
  - Study Site, Torun
  - Study Site, Wroclaw
- Romania (5):
  - Study Site, Cluj-Napoca, Cluj
  - Study Site, Timișoara, Timiș County
  - Study Site, Bucharest
  - Study Site, Craiova, Dolj
  - Study Site, Iași
- Russia (13):
  - Study Site, Nizhny Novgorod, Russian Federation
  - Study Site, Novosibirsk, Russian Federation
  - Study Site, Tonnelnyi Township, Russian Federation
  - Study Site, Kazan'
  - Study Site, Lipetsk
  - Study Site, Moscow
  - Study Site, Orenburg Region
  - Study Site, Petrozavodsk
  - Study Site, Saint Petersburg
  - Study Site, Saratov
  - Study Site, Tomsk
  - Study Site, Yaroslavl
  - Study Site, Yekaterinburg
- Serbia (3):
  - Study Site 1, Belgrade
  - Study Site 2, Belgrade
  - Study Site, Novi Sad
- Study Site, Taipei, Taiwan
- Ukraine (11):
  - Study Site, Dnipro
  - Study Site, Donetsk
  - Study Site 1, Kharkiv
  - Study Site 2, Kharkiv
  - Study Site, Kherson
  - Study Site, Luhansk
  - Study Site, Lviv
  - Study Site, Odesa
  - Study Site, Simferopol Crimea
  - Study Site, Temopil
  - Study Site, Vinnytsia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 524 participants at 118 trial sites in the following 13 countries: Bulgaria, Croatia, Hungary, India, Malaysia, Philippines, Poland, Romania, Russia, Serbia, Taiwan, Ukraine, and the United States.
Pre-assignment Details: 524 participants entered this trial (297 participants in the conversion phase and 510 participants in the open-label treatment phase). In the latter, 362 were de novo participants (283 participants entered into the conversion phase) and 148 rolled over from Trial NCT01149655.
Groups:
- Conversion Phase: Participants who entered this phase were converted from his or her antipsychotic to the minimum target dose of 10 mg/day aripiprazole monotherapy and continued to increase the dose up to a maximum of 30 mg/day, or for tolerability reasons, to reduce the aripiprazole dose to no less than 5 mg/day.
- Open-label Treatment Phase: Participants who entered this phase had received oral aripiprazole at a target dose of 10 to 30 mg/day, with a minimum dose of 5 mg/day, based on individual participant's response and tolerability considerations.
Period: Period 1 - Conversion Phase
Arm/Group | Conversion Phase | Open-label Treatment Phase
Started | 297 | 0
Completed | 283 | 0
Not Completed | 14 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Met Withdrawal Criteria | 1 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 7 | 0
Not completed — Protocol Deviation | 1 | 0
Period: Period 2- Open-label Treatment Phase
Arm/Group | Conversion Phase | Open-label Treatment Phase
Started | 0 | 510 (362 were de novo participants and 148 had rolled over from study NCT01149655.)
Completed | 0 | 198 (De novo participants who completed Month 24 visit or rolled over from study NCT01149655.)
Not Completed | 0 | 312
Not completed — Lost to Follow-up | 0 | 21
Not completed — Adverse Event | 0 | 33
Not completed — Sponsor Discontinued Trial | 0 | 165
Not completed — Met Withdrawal Criteria | 0 | 9
Not completed — Physician Decision | 0 | 12
Not completed — Withdrawal by Subject | 0 | 65
Not completed — Lack of Efficacy | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who entered open-label treatment phase had received oral aripiprazole at a target dose of 10 to 30 mg/day, with a minimum dose of 5 mg/day, based on individual participant's response and tolerability considerations.
Arm/Group | All Study Participants
Number analyzed (Participants) | 524
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.2 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 316
  Male | 208

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant or participant enrolled in a clinical trial and which did not necessarily have a causal relationship with the study medication. A treatment emergent adverse event (TEAE) was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study medication, whether or not considered to have a causal relationship with the study medication. A serious-AE or reaction was any untoward occurrence that, at any dose, was fatal, life-threatening, required inpatient hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was any other medically significant event that, based on appropriate medical judgment, may have jeopardized the participant and may have required medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Adverse events were recorded from the time of the informed consent was signed throughout the 24 month treatment period until the follow-up visit 30 (± 3) days after the end of trial.
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Number; unit: Participants
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 510
Participants
  Participants with TEAEs | 349
  Participants with serious TEAEs | 49
  Participants with severe TEAEs | 33
  Discontinued due to AEs | 32

2. Secondary Outcome: Incidence of Laboratory Values of Potential Clinical Relevance
Description: The laboratory values were one of the parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal values in serum chemistry, hematology, urinalyses and prolactin tests that were identified based on pre-defined criteria. Abnormal laboratory values in participants were reported as SAE/AEs and are reported in the SAE/other AE section of this report.
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Number; unit: participants
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 510
participants
  Chemistry-Alanine transaminase | 11
  Chemistry-Aspartate transaminase | 8
  Chemistry-Bilirubin, total | 20
  Chemistry-Calcium | 30
  Chemistry-Chloride | 158
  Chemistry-Cholesterol, total, fasting | 68
  Chemistry-Creatine phosphokinase, total | 40
  Chemistry-Glutamyl transferase | 78
  Chemistry-HDL cholesterol, fasting | 128
  Chemistry-LDL cholesterol, calculation, | 2
  Chemistry-Phosphorus inorganic | 135
  Chemistry-Protein, total serum | 81
  Chemistry-Triglycerides, fasting | 46
  Hematology-Eosinophils | 19
  Hematology-Hemoglobin | 14
  Hematology-White blood cell count | 9
  Urinalysis-Protein, urine | 348
  Urinalysis-Specific gravity | 188
  Others-Insulin | 49
  Others-Insulin, fasting | 78
  Others-Prolactin | 324

3. Secondary Outcome: Incidence of Physical Examination Findings of Potential Clinical Relevance
Description: The physical examination evaluation was one of the parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal changes in the following body systems: head, ears, eyes, nose, and throat; thorax; abdomen; urogenital; extremities; neurological; and skin and mucosae.
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole. Any clinically relevant abnormal changes were recorded as TEAEs.
Measure: Number; unit: participants
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 510
participants | 0

4. Secondary Outcome: Incidence of Vital Signs of Potential Clinical Relevance
Description: Vital signs are taken at Baseline, Weeks 1, 2, 3, 4, 6, 8, and Months 3, 4, 6, 9, 12, 15, 18, 21, 24 of Phase 2 (Visits beyond Month 12 only for de novo subjects). Assessments included orthostatic (supine and standing) blood pressure (BP), heart rate and body temperature. Incidence of TEAEs of potential clinical relevance included abnormal values in heart rate, systolic and diastolic blood pressure, respiratory rate and weight that were identified based on pre-defined criteria. Abnormal vital signs in participants were reported as SAE/AEs and are reported in the SAE/other AE section of this report.
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Number; unit: participants
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 510
participants
  Heart rate supine-Increase ≥15 bpm | 1
  Heart rate supine-Decrease ≥15 bpm | 1
  Heart rate standing-Increase ≥15 bpm | 4
  Heart rate standing-Decrease ≥15 bpm | 0
  Systolic supine bp-Increase ≥20 mmHg | 36
  Systolic supine bp-Decrease ≥20 mmHg | 31
  Systolic standing bp-Increase ≥20 mmHg | 38
  Systolic standing bp-Decrease ≥20 mmHg | 40
  Diastolic supine bp-Increase ≥15 mmHg | 41
  Diastolic supine bp-Decrease ≥15 mmHg | 19
  Diastolic standing bp-Increase ≥15 mmHg | 53
  Diastolic standing bp-Decrease ≥15 mmHg | 13
  Weight gain ≥7% | 195
  Weight loss ≥7% | 45

5. Secondary Outcome: Mean Change From Baseline by Week in Abnormal Involuntary Movement Scale (AIMS)
Description: The AIMS Scale was an extrapyramidal symptoms (EPS) rating scale. The AIMS is a 12 item scale. The first 10 items e.g. facial and oral movements (items 1-4), extremity movements (items 5 and 6), trunk movements (item 7), investigators global assessment of dyskinesia (items 8 to 10). The first 10 items are rated from 0 to 4 (0=best, 4=worst). Items 11 and 12, related to dental status, have dichotomous responses, 0=no and 1=yes. The AIMS Total Score is the sum of the ratings for the first seven items. The possible total scores are from 0 to 28.
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 510
Units on a scale
  Week 1 (N=486) | -0.02 (0.24)
  Week 2 (N=507) | -0.01 (0.25)
  Week 3 (N=507) | 0.01 (0.36)
  Week 4 (N=507) | -0.01 (0.27)
  Week 6 (N=507) | 0.02 (0.56)
  Week 8 (N=507) | -0.02 (0.28)
  Month 3 (N=507) | -0.00 (0.31)
  Month 6 (N=507) | -0.02 (0.40)
  Month 9 (N=506) | 0.01 (0.55)
  Month 12 (N=507) | -0.02 (0.41)
  Month 15 (N=360) | -0.01 (0.43)
  Month 18 (N=360) | -0.04 (0.35)
  Month 21 (N=360) | -0.01 (0.52)
  Month 24 (N=360) | -0.04 (0.34)

6. Secondary Outcome: Mean Change From Baseline by Week in Simpson-Angus Scale (SAS) Total Score
Description: The SAS is a rating scale used to measure EPS. The SAS scale consists of a list of 10 symptoms of parkinsonism (gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, head rotation, glabella tap, tremor, salivation, and akathisia), with each item rated from 0 to 4, with 0 being normal and 4 being the worst. The SAS Total score is sum of ratings for all 10 items, with possible Total scores from 0 to 40.
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 510
Units on a scale
  Week 1 (N=486) | -0.08 (0.89)
  Week 2 (N=507) | -0.11 (1.22)
  Week 3 (N=507) | -0.08 (1.23)
  Week 4 (N=507) | -0.18 (1.37)
  Week 6 (N=507) | -0.12 (1.49)
  Week 8 (N=507) | -0.21 (1.34)
  Month 3 (N=507) | -0.23 (1.56)
  Month 6 (N=507) | -0.31 (1.48)
  Month 9 (N=506) | -0.35 (1.50)
  Month 12 (N=507) | -0.36 (1.51)
  Month 15 (N=360) | -0.43 (1.78)
  Month 18 (N=360) | -0.48 (1.74)
  Month 21 (N=360) | -0.49 (1.82)
  Month 24 (N=360) | -0.53 (1.81)

7. Secondary Outcome: Mean Change From Baseline by Week in Barnes Akathisia Rating Scale (BARS) Score
Description: The BARS was an EPS rating scale. The BARS was used to assess the presence and severity of akathisia. This scale consists of 4 items. Only the 4th item, the Global Clinical Assessment of Akathisia, was evaluated in this trial. This item is rated on a 6 point scale, with 0 being best (absent) and 5 being worst (severe akathisia).
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 510
Units on a scale
  Week 1 (N=487) | -0.02 (0.26)
  Week 2 (N=507) | -0.02 (0.35)
  Week 3 (N=507) | -0.02 (0.35)
  Week 4 (N=507) | -0.03 (0.33)
  Week 6 (N=507) | -0.03 (0.36)
  Week 8 (N=507) | -0.02 (0.41)
  Month 3 (N=507) | -0.00 (0.45)
  Month 6 (N=507) | -0.03 (0.44)
  Month 9 (N=506) | -0.04 (0.43)
  Month 12 (N=507) | -0.04 (0.42)
  Month 15 (N=360) | -0.02 (0.47)
  Month 18 (N=360) | -0.05 (0.48)
  Month 21 (N=360) | -0.04 (0.50)
  Month 24 (N=360) | -0.05 (0.47)

8. Secondary Outcome: Number of Participants With Cognitive Impairment for Each New York Assessment for Adverse Cognitive Effects of Neuropsychiatric Treatment (NY-AACENT)
Description: The NY-AACENT is not a validated scale. It was included in this trial because of concerns that regulatory authorities (the European Committee for Medicinal Products for Human Use [CHMP] and the Paediatric Sub-Committee of the European Medicinal Agency [PDCO]) had regarding drug induced cognitive impairment. No validated scale addressing these issues was available at the time of the trial. The NY-AACENT was used to detect changes in cognitive function subsequent to pharmacological or similar treatments for neurological or psychiatric problems. It was specifically designed to be used in pediatric populations (ages 12 to 17), but could have been utilized with other age groups, as appropriate.
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Number; unit: participants
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 510
participants
  Working memory | 237
  Attention/vigilance | 306
  Verbal learning/memory | 233
  Visual learning/memory | 138
  Reasoning and problem solving | 308
  Speed of processing | 276
  Social congnition | 307

9. Secondary Outcome: Baseline and Post-Baseline Tanner Staging
Description: Tanner staging was completed together with the physical examination by the same trial-affiliated clinician in the most inconspicuous manner for the participant as possible. Tanner staging assessment consisted of 2 domains (pubic hair and breast development) for girls and 3 domains (pubic hair, penis development, and testes development) for boys. A participant who reached Stage 5 (both in pubic hair and genitalia) did not need to continue with Tanner Staging assessment and the Tanner Staging scales of this participant were imputed as 5 for all of the following scheduled time points up to and including the completion visit/ET visit. The clinician arrived at a single score summarizing the domains (not individual domain scores) when evaluating the participant. The total shift data for last visit is presented below.
Time Frame: Baseline to Last Visit
Population: All those participants who had received at least one dose of oral aripiprazole during the open-label treatment phase.
Measure: Number; unit: participants
Groups:
- Tanner Score at Baseline of 1; Tanner Score at Baseline of 2; Tanner Score at Baseline of 3; Tanner Score at Baseline of 4; Tanner Score at Baseline of 5: Participants who entered this phase had received oral aripiprazole at a target dose of 10 to 30 mg/day, with a minimum dose of 5 mg/day, based on individual participant's response and tolerability considerations.
Arm/Group | Tanner Score at Baseline of 1 | Tanner Score at Baseline of 2 | Tanner Score at Baseline of 3 | Tanner Score at Baseline of 4 | Tanner Score at Baseline of 5
Number analyzed (Participants) | 7 | 24 | 79 | 196 | 204
participants
  Last Visit (Post-Baseline score of 1) (N= 1) | 1 | 0 | 0 | 0 | 0
  Last Visit (Post-Baseline score of 2) (N= 9) | 4 | 5 | 0 | 0 | 0
  Last Visit (Post-Baseline score of 3) (N= 39) | 2 | 9 | 28 | 0 | 0
  Last Visit (Post-Baseline score of 4) (N= 134) | 0 | 7 | 33 | 94 | 0
  Last Visit (Post-Baseline score of 5) (N= 327) | 0 | 3 | 18 | 102 | 204

10. Secondary Outcome: Mean Change From Baseline for Columbia-Suicide Severity Rating Scale (C-SSRS) in Suicidal Ideation Intensity Total Score
Description: Suicidality was defined as reporting at least one occurrence of any suicidal behavior or suicidal ideation. Suicidal behavior was defined as reporting any type of suicidal behaviors (actual attempt, interrupted attempt, aborted attempt, and preparatory acts or behavior). Suicidal ideation was defined as reporting any type of suicidal ideation. The suicidal ideation intensity total score is the sum of intensity scores of 5 items (frequency, duration, controllability, deterrents, and reasons for ideation). The score of each intensity item ranges from 0 (none) to 5 (worst) which leads to the range of the total score from 0 to 25. A missing score of any item resulted in a missing total score. If no suicidal ideation was reported, a score of 0 was given to the intensity scale.
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 510
Units on a scale
  Week 1 (N= 487) | -0.4 (2.1)
  Week 2 (N= 483) | -0.4 (2.2)
  Week 3 (N= 477) | -0.4 (2.2)
  Week 4 (N= 491) | -0.4 (2.2)
  Week 6 (N= 488) | -0.3 (2.1)
  Week 8 (N= 484) | -0.4 (2.0)
  Month 3 (N= 478) | -0.3 (2.2)
  Month 4 (N= 472) | -0.3 (2.1)
  Month 6 (N= 458) | -0.2 (2.5)
  Month 9 (N= 407) | -0.2 (1.8)
  Month 12 (N= 302) | -0.3 (2.0)
  Month 15 (N= 261) | -0.2 (1.9)
  Month 18 (N= 247) | -0.1 (2.0)
  Month 21 (N= 212) | -0.1 (1.8)
  Month 24 (N= 180) | -0.0 (1.9)
  Last Visit (N= 507) | -0.1 (2.5)

11. Secondary Outcome: Incidence of Suicidality, Suicidal Behavior and Suicidal Ideation
Description: Suicidality was defined as reporting at least one occurrence of any suicidal behavior or suicidal ideation. Suicidal behavior was defined as reporting any type of suicidal behaviors (actual attempt, interrupted attempt, aborted attempt, and preparatory acts or behavior). Suicidal ideation was defined as reporting any type of suicidal ideation. The below reported N value is the number of participants with specified suicidal ideation/behavior at the given time point.
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Number; unit: participants
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 510
participants
  Complete suicidality | 0
  Suicidality | 32
  Suicidal behavior | 5
  Emergence of suicidal behavior | 3
  Suicidal ideation | 31
  Emergence of suicidal ideation | 19
  Emergence of serious suicial ideation | 2
  Worsening of suicidal ideation | 26

12. Secondary Outcome: Percentage of Participants Who Discontinued Due to All Adverse Events
Description: The percentage of participants who discontinued due to all causes other than sponsor terminating the trial was measured from the date of entering the open-label treatment phase to the date of ET for discontinued participants in the open-label treatment phase (ie, time to discontinuation = date of discontinuation [or date of completion for completed participants] - date of participant entering the open-label treatment phase + 1). If the participants completed the trial or were discontinued due to the sponsor terminating the trial, they were censored at the time of completion or trial termination, respectively.
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 510
percentage of participants
  From study NCT01149655 (N= 148) | 3.4
  De Novo (N= 362) | 7.7

13. Secondary Outcome: Mean Change From Baseline in Positive and Negative Symptoms Score (PANSS) Total Score
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS total score was the sum of the rating scores for 7 positive scale items, 7 negative scale items, and 16 general psychopathology scale items from the PANSS panel. The PANSS total score ranged from 30 (best possible outcome) to 210 (worst possible outcome).
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 510
Units on a scale
  Month 12 (N= 414) | -9.98 (14.66)
  Month 24 (N= 267) | -12.52 (15.70)

14. Secondary Outcome: Mean Change From Baseline in PANSS Positive Subscale Score
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS positive subscale score was the sum of the rating scores for the 7 positive scale items from the PANSS panel. The 7 positive symptom constructs are delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. The PANSS Positive Subscale ranges from 7 (absence of symptoms) to 49 (extremely severe symptoms).
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 510
Units on a scale
  Month 12 (N= 414) | -2.57 (4.96)
  Month 24 (N= 267) | -2.91 (5.13)

15. Secondary Outcome: Mean Change From Baseline in PANSS Negative Subscale Score
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS negative subscale score was the sum of the rating scores for the 7 negative scale items from the PANSS panel. The 7 negative symptom constructs: blunted affect, emotional withdrawal, poor rapport, passive apathetic withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. The PANSS Negative Subscale ranges from 7 (absence of symptoms) to 49 (extremely severe symptoms).
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 510
Units on a scale
  Month 12 (N= 414) | -2.79 (4.17)
  Month 24 (N= 267) | -3.48 (4.63)

16. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score
Description: The severity of illness for each participant was rated using the CGI-S scale. To assess CGI-S, the study physician answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0 = not assessed; 1 = normal, not ill at all; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 510
Units on a scale
  Month 12 (N= 414) | -0.66 (0.96)
  Month 24 (N= 267) | -0.77 (1.04)

17. Secondary Outcome: Mean Change in Clinical Global Impression-Improvement (CGI-I) Score
Description: The efficacy of trial medication were rated for each participant using the CGI-I scale. The study physician must rate the participant's total improvement whether or not it is due entirely to drug treatment. All responses were compared to the participant's condition at baseline. Response choices include: 0 = not assessed; 1 =very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 =minimally worse; 6 = much worse; and 7 = very much worse.
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 510
Units on a scale
  Month 12 (N= 408) | 2.62 (1.16)
  Month 24 (N= 263) | 2.38 (1.15)

18. Secondary Outcome: Mean Change From Baseline in Young Mania Rating Scale (YMRS) Score
Description: The YMRS consists of 11 items assessing the core symptoms of mania and was used to assess participants with bipolar I disorder, manic and mixed episodes with or without psychotic features: elevated mood, increased motor activity - energy, sexual interest, sleep, irritability, speech (rate and amount), language - thought disorder, content, disruptive - aggressive behavior, appearance, and insight. Each item had 5 or 9 grades of severity, with lower scores indicating milder symptoms. The number of raters within each trial center was to be kept to a minimum. The YMRS Total Score (range 0 to 44) is the sum of the rating scores for 11 items for assessing the core symptoms of mania. A missing value for any YMRS assessment item(s) could have resulted in a missing YMRS Total Score. A higher YMRS Total Score represents greater severity. In this study, 94 participants had bipolar disorder, this explains the N=94 in the table below and these were de novo participants.
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 94
Units on a scale
  Month 12 (N= 93) | -9.71 (10.23)
  Month 24 (N= 93) | -10.02 (10.21)

19. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression Scale - Bipolar (CGI-BP) Version Severity Score
Description: The CGI-BP scale refers to the global impression of the subject with respect to bipolar disorder. The scale rated the subject's Severity of Illness (CGI-BP-Severity: mania, depression, and overall bipolar illness) and Change From Preceding Phase (CGI-BP-Improvement: mania, depression, and overall bipolar illness) based on a 7- or 8-point scale. Severity of Illness (CGI-BP-Severity) was rated at all visits. At each visit other than Day 0 (Baseline), the Change From Preceding Phase (CGI-BP-Improvement) was judged with respect to participant's condition at Baseline. The CGI-BP Severity Scores (range 1 to 7), as well as CGI-BP Improvement Scores (range 1 to 7) are single-item rating scores, with higher scores representing greater severity or less improvement. Data for 94 de novo participants were available with bipolar disorder.
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 94
Units on a scale
  Month 12 (N= 93) | -1.26 (1.33)
  Month 24 (N= 93) | -1.30 (1.37)

20. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression Scale - Bipolar Version Improvement Score
Description: The CGI-BP scale refers to the global impression of the subject with respect to bipolar disorder. The scale rated the subject's Severity of Illness (CGI-BP-Severity: mania, depression, and overall bipolar illness) and Change From Preceding Phase (CGI-BP-Improvement: mania, depression, and overall bipolar illness) based on a 7- or 8-point scale. Severity of Illness (CGI-BP-Severity) was rated at all visits. At each visit other than Day 0 (Baseline), the Change From Preceding Phase (CGI-BP-Improvement) was judged with respect to participant's condition at Baseline. The CGI-BP Severity Scores (range 1 to 7), as well as CGI-BP Improvement Scores (range 1 to 7) are single-item rating scores, with higher scores representing greater severity or less improvement. Only 94 participants had data at Baseline to explain the N=94 in the table below and these were de novo participants.
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 94
Units on a scale
  Month 12 (N= 93) | 2.27 (1.28)
  Month 24 (N= 93) | 2.17 (1.27)

21. Secondary Outcome: Mean Change From Baseline in General Behavior Inventory (GBI) Scale Total Score for Mania and Depression in Both Parent/Guardian and Subject Version of the Scale
Description: The GBI is a self-report inventory with 73 items focusing on mood-related behaviors, including depressive, hypomanic, and biphasic symptoms. For this trial, two 20-item subscales were utilized: one was completed by the parent/guardian or legal representative, as applicable for local laws, and the other was completed by the participant. Responses were given on a 4-point Likert scale, with 0 being never or hardly ever and 3 being very often or almost constantly. The GBI Total Score for mania (range 0 to 30) is the sum of scores for items 1 to 10 and the GBI Total Score for depression (range 0 to 30) is the sum of scores for items 11 to 20 in the GBI Parent/Guardian or Subject Version panel. Scores from the Parent/Guardian and participant Versions were summarized separately. A missing value for any GBI assessment items could have resulted in a missing GBI Total Score. High scores represent greater psychopathology. Data was only available for 80 de novo participants with bipolar disorder.
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 80
Units on a scale
  Month 12 (N= 78) | -1.62 (7.20)
  Month 24 (N= 78) | -1.82 (7.37)

22. Secondary Outcome: Mean Change From Baseline in the Attention Deficit Hyperactive Disorders Rating (ADHD-RS-IV) Scale Score
Description: The ADHD-RS-IV is a reliable and easy-to-administer instrument both for diagnosing ADHD in children and adolescents and for assessing treatment response. Containing 18 items, the scale was linked directly to DSM-IV-TR diagnostic criteria for ADHD. There were 3 versions of the scale: a parent questionnaire on home behaviors (English), a parent questionnaire on home behaviors (Spanish), and a teacher questionnaire on classroom behaviors. For this trial, the parent questionnaire on home behaviors (English) was utilized. The ADHD-RS-IV Total Score (range 0 to 54) is the sum of rating scores for 18 items, with higher scores representing greater severity. A missing value for any ADHD-RS-IV assessment items could have resulted in a missing ADHD-RS-IV Total Score. Data were only available for 82 participants with bipolar disorder and these were de novo participants.
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 82
Units on a scale
  Month 12 (N= 81) | -3.25 (10.43)
  Month 24 (N= 81) | -2.53 (10.73)

23. Secondary Outcome: Mean Change From Baseline in Children's Global Assessment Scale (CGAS) in Bipolar (de Novo Participants)
Description: The CGAS is a 100-point rating scale measuring psychological, social, and school functioning for children aged 6 to 17. It was adapted from the Adults Global Assessment Scale. The Global Assessment Scale was a rating scale for evaluating the overall functioning of a participant during a specified time period on a continuum from psychological or psychiatric sickness to health. The CGAS is a valid and reliable tool for rating a child's general level of functioning on a health-illness continuum. The CGAS was developed by Schaffer and colleagues to provide a global measure of severity of disturbance in children and adolescents. The CGAS Score (range 1 to 100) is a single-item score for rating a child's general level of functioning on a health-illness continuum, with higher scores representing better functioning.
Time Frame: Baseline to Month 24
Population: All participants who had received at least one dose of oral aripiprazole.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Treatment Phase
Number analyzed (Participants) | 94
Units on a scale
  Month 12 (N= 93) | 14.17 (16.01)
  Month 24 (N= 93) | 14.00 (16.23)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the signing of the informed consent, during the 24-month treatment period until the follow-up visit 30 (± 3) days after the end of trial.
Groups:
- Conversion Phase: Participants who entered this phase were converted from his or her antipsychotic to the minimum target dose of 10 mg/day aripiprazole monotherapy and continue to increase the dose up to a maximum of 30 mg/day, or for tolerability reasons, to reduce the aripiprazole dose to no less than 5 mg/day.
Arm/Group | Conversion Phase | Open-label Treatment Phase
Serious Adverse Events (participants affected / at risk) | 2/297 | 49/510
Other Adverse Events (participants affected / at risk) | 40/297 | 194/510
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conversion Phase (N=297) | Open-label Treatment Phase (N=510)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Irritability (General disorders) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Blood creatine phosphokinase (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 18
Suicidal ideation (Psychiatric disorders) | 0 | 8
Bipolar disorder (Psychiatric disorders) | 0 | 7
Aggression (Psychiatric disorders) | 0 | 3
Agitation (Psychiatric disorders) | 0 | 3
Hallucination, auditory (Psychiatric disorders) | 0 | 2
Suicide attempt (Psychiatric disorders) | 0 | 2
Bipolar I disorder (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Self injurious behaviour (Psychiatric disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Conversion Phase (N=297) | Open-label Treatment Phase (N=510)
Vomiting (Gastrointestinal disorders) | 4 | 30
Nasopharyngitis (Infections and infestations) | 5 | 34
Weight increased (Investigations) | 1 | 38
Headache (Nervous system disorders) | 23 | 67
Somnolence (Nervous system disorders) | 20 | 33
Anxiety (Psychiatric disorders) | 6 | 32
Schizophrenia (Psychiatric disorders) | 1 | 30

LIMITATIONS AND CAVEATS:
The study was terminated by the Sponsor as the European Medicines Agency P/99/2011Aripiprazole PIP which directed the sponsor to provide 2 years of safety data for at least 100 participants. The objective was met in April 2014.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No